CLINICAL TRIAL: NCT02880605
Title: Validation of Chinese Version Appropriate Use Criteria for Coronary Revascularization
Status: Completed | Type: Observational
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2016-1-4031
Record Dates: First submitted 2016-08-16; First posted 2016-08-26 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Appropriate Use Criteria; Coronary Revascularization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- appropriate in appropriate indications
- inappropriate in appropriate indications
- appropriate in inappropriate indications
- inappropriate in inappropriate indications

SUMMARY:
Coronary revascularization (CR) is increasing rapidly in China and varies significantly in proportion ( PCI:CABG=15:1). Few studies assess the appropriateness of CR in China. Recently, National Center for Cardiovascular Disease organized experts to release Chinese version appropriate use criteria(C-AUC) for coronary revascularization by RAND method aimed at regulating indications of CR. The criteria is considered to contribute to clinical practices, quality assessment and health insurance policy, however, the validation of C-AUC is unknown.

Thus the investigators study aims at assessing the validation of Chinese AUC by multi-center prospective registry. The investigators will recruit 4000 patients undergoing elective coronary angiography with positive outcome consecutively and collect baseline information. Sequently, one-year follow up will be done to collect the prognose, including death, rehospitalization, medicine, medical compliance and life quality etc. One hand, the investigators will compare the outcomes between different therapies in the same indications according to C-AUC to evaluate the validation of C-AUC. On the other hand, the investigators will evaluate the rationality of CAD therapy in Beijing by C-AUC.

ELIGIBILITY:
Inclusion Criteria:

* Undergo elective coronary angiography in department of cardiology in period of study
* Written informed consent

Exclusion Criteria:

* Age ≤18 years of age
* Illiteracy, vision/audition disorder, cognitive disorder etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergo elective coronary angiography in department of cardiology in period of study.
  Patients are written informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 11235 (Actual)
Dates: Start 2016-08; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 1 year
  death, nonfatal myocardial infarction, cerebrovascular event, repeat revascularization

SECONDARY OUTCOMES:
death | 1 year
recurrent hospitalizations for acute coronary syndrome (ACS) | 1 year
cerebrovascular event | 1 year
repeat revascularization | 1 year
cost for hospitalization | 1 year
  Total cost of hospitalization and rehospitalization for cardiac disease in follow-up time

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin S, Zhang H, Chen SP, Rao CF, Wu F, Zhou FJ, Wang Y, Yan HB, Dou KF, Wu YJ, Tang YD, Xie LH, Guan CD, Xu B, Zheng Z. Mis-estimation of coronary lesions and rectification by SYNTAX score feedback for coronary revascularization appropriateness. Chin Med J (Engl). 2020 Jun 5;133(11):1276-1284. doi: 10.1097/CM9.0000000000000827. PMID 32452896
- [Derived] Lin S, Zhang H, Rao CF, Chen SP, Qiao SB, Yan HB, Dou KF, Wu YJ, Tang YD, Yang XC, Shen ZJ, Liu J, Zheng Z; Beijing Coronary Angiography Registry Collaborative Group. Assessing the association of appropriateness of coronary revascularization and 1-year clinical outcomes for patients with stable coronary artery disease in China. Chin Med J (Engl). 2020 Jan 5;133(1):1-8. doi: 10.1097/CM9.0000000000000592. PMID 31923098